CLINICAL TRIAL: NCT00020553
Title: We Can Cope: Family Support When A Parent Has Cancer
Brief Title: Video Support Program For Families With a Parent Newly Diagnosed With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inflexxion, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000068602; INFLEXXION-000080; ITS-000080; NCI-V01-1659
Record Dates: First submitted 2001-07-11; First posted 2004-02-16 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2006-10

CONDITIONS: Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment
MeSH Terms: interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: A videotape support program may help families improve communication and coping skills when a parent is diagnosed with cancer.

PURPOSE: Randomized trial to study the effectiveness of a video support program for families who have a parent who has been newly diagnosed with cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine if families who participate in a video support program function better as a family in the areas of communication, togetherness, and overall increased ability to cope when a parent is newly diagnosed with cancer. II. Determine if participation in this program decreases stress-related illness in the well members of the family. III. Determine the safety of this program. IV. Determine patient/family and medical provider satisfaction with this program.

OUTLINE: This a randomized study. Adult parent participants and spouses undergo a baseline assessment over approximately 1 hour comprising completion of a self-assessment form followed by an interview. Families are then randomized to one of two arms. Arm I: Adult parent participants receive a video support program comprising 3 videotapes (parent tape, adolescent tape, and child tape) and a parent guidebook. The parents are encouraged to screen the videotapes and decide whether to have their child and/or adolescent view the program. Arm II: Adult parent participants receive no video support material. Families may view the video program after study completion. Adult parent participants in both arms complete follow-up assessments at 6 and 12 weeks. This clinical trial is being conducted at the locations listed below. If you are interested in this clinical trial but unable to visit these locations, please call #1-800-848-3895 ext. 226 and ask for more information about the We Can Cope study.

PROJECTED ACCRUAL: A total of 230 families will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Parent with a first diagnosis of cancer within the past 5 years No recurrence of a previously diagnosed cancer Must have at least 1 child between the ages of 6 and 18 Ill parent must live with child/children at least 50% of the time No plans to move out-of-state within the next 3 months

PATIENT CHARACTERISTICS: Age: See Disease Characteristics Any age Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No psychotic disorder (such as schizophrenia) or a brain/psychiatric disorder due to disease/illness

PRIOR CONCURRENT THERAPY: Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-08

CONTACTS AND LOCATIONS:
Overall Officials: Jonas I. Bromberg, Study Chair — Inflexxion, Inc.
Locations (5):
- United States (5):
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - Inflexxion, Newton, Massachusetts
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Buddy Kemp Caring House, Charlotte, North Carolina
  - Baylor University Medical Center, Dallas, Texas